CLINICAL TRIAL: NCT07313228
Title: Pulsed Field Ablation of Non-valvular Atrial Fibrillation After Left Atrial Appendage Occlusion: A Prospective, Single-center, Single-arm Clinical Trial
Brief Title: Pulsed Field Ablation for Non-valvular Atrial Fibrillation After Left Atrial Appendage Occlusion
Acronym: PFA after LAAO
Status: Not yet recruiting | Type: Observational
Sponsor: First Affiliated Hospital of Ningbo University (Network)
Responsible Party: Sponsor
Other Study IDs: NBUFH-2025Y-289A; MR-33-25-078136 (Other: Medical Research Registration and Record Information System)
Record Dates: First submitted 2025-12-17; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Atrial Fibrillation; Left Atrial Appendage Occlusion; Pulsed Field Ablation
Keywords: Atrial Fibrillation; left atrial appendage occlusion; pulsed field ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PFA after LAAO group: The patients in this group have previously undergone Left Atrial Appendage Occlusion (LAAO) surgery and are scheduled to undergo Pulsed Field Ablation (PFA). The study will only collect comprehensive data throughout their treatment process without introducing any additional interventions.
  Interventions: Procedure: Pulsed Field Ablation

INTERVENTIONS:
Procedure: Pulsed Field Ablation — Pulsed Field Ablation is a surgical technique for atrial fibrillation ablation that uses pulsed electric fields.

SUMMARY:
This is a single-center, prospective, single-arm clinical trial designed to evaluate the safety and efficacy of pulsed field ablation (PFA) after left atrial appendage occlusion (LAAO) in patients with non-valvular atrial fibrillation (AF). The trial will include patients who have undergone successful LAAO and have symptomatic AF that is refractory to or intolerant of class I or III antiarrhythmic drugs. The primary objective is to assess the effectiveness of PFA in preventing AF recurrence and its safety, including the occurrence of serious adverse events. Patients will be followed up for 12 months post-procedure to evaluate outcomes such as recurrence of AF, complications, and device-related issues.

DETAILED DESCRIPTION:
This clinical trial aims to explore the safety and efficacy of pulsed field ablation (PFA) in patients who have undergone left atrial appendage occlusion (LAAO) for the treatment of non-valvular atrial fibrillation (AF). LAAO is an effective strategy for stroke prevention in patients with AF, and PFA is a novel non-thermal ablation technique that may offer advantages over traditional radiofrequency ablation, particularly by minimizing collateral damage to surrounding structures.

The study will enroll adult patients aged 18-75 years who have symptomatic AF that is refractory to or intolerant of at least one class I or III antiarrhythmic drug and have previously undergone LAAO. The trial will be conducted at a single center, with each participant receiving PFA after LAAO.

The procedure will involve the use of PFA to ablate the left atrium and achieve electrical isolation of the pulmonary veins, guided by fluoroscopy and intracardiac echocardiography. The primary endpoint is the absence of any atrial arrhythmia (AF or atrial flutter) over a 12-month follow-up period, assessed via ECG and Holter monitoring. Secondary endpoints include acute procedural success (i.e., achieving pulmonary vein isolation), as well as the assessment of complications such as phrenic nerve injury, device-related issues, and other adverse events.

The study will monitor patients closely post-procedure at 24 hours, 1 month, 3 months, 6 months, and 12 months, assessing clinical outcomes such as recurrence of AF, device-related complications, and changes in the left atrial appendage closure device position or leak. Data from baseline evaluations, including echocardiography, CT, and blood tests, will be collected and used for comparative analysis throughout the study.

This research is expected to contribute valuable evidence on the feasibility, safety, and efficacy of combining LAAO with PFA in the treatment of non-valvular AF, potentially benefiting a large population of patients who have limited treatment options.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-75 years;
2. Documented symptomatic atrial fibrillation;
3. Ineffective or intolerant to at least one class I or III antiarrhythmic drug;
4. Able to fully understand the treatment protocol, voluntarily sign the informed consent form, and willing to undergo the required examinations, procedures, and follow-up.

Exclusion Criteria:

1. Patients who have previously undergone left atrial surgery;
2. Left atrial thrombus;
3. Patients with pulmonary agenesis;
4. Female patients of reproductive age who cannot use effective contraception within 12 months after enrollment;
5. Left atrial anteroposterior diameter ≥ 55 mm;
6. Left ventricular ejection fraction (LVEF) ≤ 40%;
7. Patients who have previously undergone interatrial septal repair or removal of atrial myxoma;
8. Patients with active implanted devices (e.g., pacemaker, ICD);
9. Patients with NYHA heart failure class III-IV;
10. Patients with a clear history of cerebrovascular disease (including cerebral hemorrhage, stroke, or TIA) within the past 6 months;
11. Patients who have experienced cardiovascular events (e.g., acute myocardial infarction, coronary intervention or bypass surgery, valve replacement or repair, atrial or ventricular surgery) within the past 3 months;
12. Patients with acute or severe systemic infections;
13. Patients with severe liver or kidney disease, malignancy, or end-stage disease that may affect the treatment, assessment, or compliance of the trial (as judged by the investigator);
14. Patients with significant bleeding tendency, hypercoagulable state, or severe hematologic disorders;
15. Patients who have participated or are currently participating in another clinical trial within the past 12 months prior to enrollment;
16. Patients who the investigator deems unsuitable for participation in this trial.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The selected population consists of adult patients with a documented history of atrial fibrillation who have undergone left atrial appendage occlusion and are planned to undergo pulsed field ablation due to ineffective drug treatment. Additionally, they must not have any surgical contraindications.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
No recurrence of atrial arrhythmias within 12 months | 12month
  Defined as the absence of such arrhythmias in the efficacy evaluation period (from blanking period to the end of 12-month follow-up) based on ECG data (including both surface ECG and 24-hour Holter monitoring).

SECONDARY OUTCOMES:
Ablation success | Instantly
  Defined as the maintenance of electrical isolation of the pulmonary veins, regardless of whether isoproterenol is used, after programmed stimulation.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Blackshear JL, Odell JA. Appendage obliteration to reduce stroke in cardiac surgical patients with atrial fibrillation. Ann Thorac Surg. 1996 Feb;61(2):755-9. doi: 10.1016/0003-4975(95)00887-X. PMID 8572814
- [Background] Reddy VY, Doshi SK, Kar S, Gibson DN, Price MJ, Huber K, Horton RP, Buchbinder M, Neuzil P, Gordon NT, Holmes DR Jr; PREVAIL and PROTECT AF Investigators. 5-Year Outcomes After Left Atrial Appendage Closure: From the PREVAIL and PROTECT AF Trials. J Am Coll Cardiol. 2017 Dec 19;70(24):2964-2975. doi: 10.1016/j.jacc.2017.10.021. Epub 2017 Nov 4. PMID 29103847
- [Background] Osmancik P, Herman D, Neuzil P, Hala P, Taborsky M, Kala P, Poloczek M, Stasek J, Haman L, Branny M, Chovancik J, Cervinka P, Holy J, Kovarnik T, Zemanek D, Havranek S, Vancura V, Opatrny J, Peichl P, Tousek P, Lekesova V, Jarkovsky J, Novackova M, Benesova K, Widimsky P, Reddy VY; PRAGUE-17 Trial Investigators. Left Atrial Appendage Closure Versus Direct Oral Anticoagulants in High-Risk Patients With Atrial Fibrillation. J Am Coll Cardiol. 2020 Jun 30;75(25):3122-3135. doi: 10.1016/j.jacc.2020.04.067. PMID 32586585
- [Background] Tam MTK, Kojodjojo P, Lam YY, Chow J, Wong C, Kam KK, Wong GLN, Chan CP, Chan JYS, So KC. Combined pulsed field ablation and left atrial appendage occlusion: A multicenter comparative study. Heart Rhythm. 2025 Oct;22(10):2579-2584. doi: 10.1016/j.hrthm.2025.03.1968. Epub 2025 Mar 21. PMID 40122196
- [Background] Beney J, Galea R, Siontis G, Grani C, Kueffer T, Brugger N, Reichlin T, Raber L, Roten L. Feasibility study on atrial fibrillation ablation with pulsed field ablation and concomitant occlusion of the left atrial appendage. Europace. 2024 Jul 2;26(7):euae176. doi: 10.1093/europace/euae176. PMID 38917059